CLINICAL TRIAL: NCT01924559
Title: Comparison of Airway Intubation Devices When Using a Biohazard Suit: A Feasibility Study
Brief Title: Comparison of Airway Intubation Devices When Using a Biohazard Suit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Marna Rayl Greenberg, Director of Emergency Medicine Research, Lehigh Valley Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00000982
Record Dates: First submitted 2013-08-06; First posted 2013-08-16 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Intubation; Difficult
Keywords: Airway

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Direct Laryngoscopy & standard clothing (Active Comparator): Residents will intubate manikin using DL while wearing standard clothing.
  Interventions: Other: standard clothing; Device: Direct Laryngoscopy
- Direct Laryngoscopy & Biohazard Gear (Active Comparator): Residents will intubate manikins using DL while in Biohazard gear.
  Interventions: Other: Biohazard gear; Device: Direct Laryngoscopy
- Glidescope & standard clothing (Experimental): Residents will intubate manikins using Glidescope while wearing standard clothing.
  Interventions: Other: standard clothing; Device: Glidescope
- Glidescope & Biohazard Gear (Active Comparator): Residents will intubate manikins using Glidescope while wearing Biohazard gear.
  Interventions: Other: Biohazard gear; Device: Glidescope
- Supraglottic Airway & standard clothing (Active Comparator): Residents will intubate manikins using Supraglottic Airway while wearing standard clothing.
  Interventions: Other: standard clothing; Device: Supraglottic Airway
- Supraglottic Airway and Biohazard gear (Active Comparator): Residents will intubate manikins using Supraglottic airway while wearing biohazard gear.
  Interventions: Other: Biohazard gear; Device: Supraglottic Airway

INTERVENTIONS:
Other: standard clothing
  Arms: Direct Laryngoscopy & standard clothing; Glidescope & standard clothing; Supraglottic Airway & standard clothing
Other: Biohazard gear
  Arms: Direct Laryngoscopy & Biohazard Gear; Glidescope & Biohazard Gear; Supraglottic Airway and Biohazard gear
Device: Direct Laryngoscopy
  Other Names: (the classic standard of care)
  Arms: Direct Laryngoscopy & Biohazard Gear; Direct Laryngoscopy & standard clothing
Device: Glidescope
  Arms: Glidescope & Biohazard Gear; Glidescope & standard clothing
Device: Supraglottic Airway
  Other Names: Supraglottic Airway Laryngopharyngeal Tube
  Arms: Supraglottic Airway & standard clothing; Supraglottic Airway and Biohazard gear

SUMMARY:
We will investigate the impact biohazard gear has on time to successful intubation and, in particular, determine how the Supraglottic Airway Laryngopharyngeal Tube (Ecolab, Columbus, Missouri) device compares to traditional direct laryngoscopy and fiber-optic (video) intubation techniques.

DETAILED DESCRIPTION:
This study will take place in an academic/training facility at Lehigh Valley Health Network simulating intubation during a bio-terrorism attack. As a part of their usual (standard of care) residency education, the study volunteers will be participating in a day-long airway training course in the Fall of 2013 where each of the tested devices will be introduced and the residents will be able to practice using them on a variety of training mannequins.

As part of this training, the enrolled study subjects will be timed using each of three intubation devices, both with and without wearing biohazard protective gear, for a total of six measurements per resident. Residents will have been assigned chronological numbers as they arrived and signed in for the course. These numbers will be also used for study identification numbers. Subjects will be randomized by odd or even identification numbers as to whether they will make their initial attempt in street clothing or the biohazard suit. This will help control for individual subject's skill learning. The subject will then intubate the same mannequins using each of the tested devices.

The order of devices used will be the same as in actual clinical practice: 1) Direct Laryngoscopy (the classic standard of care), 2) the GlideScope or C-MAC video laryngoscope (fiber-optic technology, which has become increasingly popular among emergency physicians), and 3) the Supraglottic Airway Laryngopharyngeal Tube airway device (an inexpensive, convenient supraglottic device that allows for a blind intubation technique through the device).

Data will be collected, per device, on the time taken and tubes used for each attempt. Demographic information will also be collected from participants such as gender, resident year, prior intubation experience, prior exposure to each of the tested devices, and experience wearing a biohazard suit. Study participants' satisfaction with each of the devices will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Medicine residents who volunteer to participate and allow their data to be used for research purposes

Exclusion Criteria:

* Not an Emergency resident who volunteers to participate and allow their data to be used for research purposes

Ages: 18 Years to 126 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lipkin, DPM, CIP, Study Director — Director, Research Participant Protection Office
Locations (1):
- Lehigh Valley Hospital, Allentown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weaver KR, Barr GC Jr, Long KR, Diaz L Jr, Ratner AS, Reboul JP, Sturm DA, Greenberg MR, Dusza SW, Glenn-Porter B, Kane BG. Comparison of airway intubation devices when using a biohazard suit: a feasibility study. Am J Emerg Med. 2015 Jun;33(6):810-4. doi: 10.1016/j.ajem.2015.02.051. Epub 2015 Mar 6. PMID 25817200

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All participants were randomized into groups testing three intubation devices while wearing standard clothing or biohazard gear..
Period: Overall Study
Arm/Group | All Study Participants
Started | 37 (All 37 participants were scored under the same six scenarios, resulting in 222 observations.)
Completed | 37 (The order in which subjects started scenarios (in biohazard gear vs street clothing) was randomized)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Prospectively enrolled EM residents, including PGY 1s through 4s; each resident was observed performing all six arms of the study.
Groups:
- SALT and Biohazard Gear: All participants were tested on three intubation devices in either standard clothing or biohazard gear.
Arm/Group | SALT and Biohazard Gear
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Time to Successful Intubation
Description: Time from initiation of intubation attempt to successful 2 breaths demonstrating lung expansion, estimated less than 1 minute
Time Frame: approximately one minute
Population: EM Residents who tested/participated in each of the six groups
Measure: Mean (Full Range); unit: seconds
Groups:
- DL & Standard Clothing: Residents will intubate manikin using DL while wearing standard clothing.
  standard clothing
  DL
- DL & Biohazard Gear: Residents will intubate manikins using DL while in Biohazard gear.
  Biohazard gear
  DL
- Glidescope & Standard Clothing: Residents will intubate manikins using Glidescope while wearing standard clothing.
  standard clothing
  Glidescope
- Glidescope & Biohazard Gear: Residents will intubate manikins using Glidescope while wearing Biohazard gear.
  Biohazard gear
  Glidescope
- SALT & Standard Clothing: Residents will intubate manikins using SALT while wearing standard clothing.
  standard clothing
  SALT
- SALT and Biohazard Gear: Residents will intubate manikins using SALT while wearing biohazard gear.
  Biohazard gear
  SALT
Arm/Group | DL & Standard Clothing | DL & Biohazard Gear | Glidescope & Standard Clothing | Glidescope & Biohazard Gear | SALT & Standard Clothing | SALT and Biohazard Gear
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
seconds | 54 [25 to 189] | 106.5 [29 to 534] | 66 [19 to 298] | 83.5 [25 to 375] | 73.5 [13 to 328] | 58.5 [20 to 168]

ADVERSE EVENTS:
Time Frame: Minimal risk study, N/A.
Description: Minimal risk study, N/A.
Groups:
- SALT and Biohazard Gear: Residents will intubate manikins using SALT while wearing biohazard gear.
  Biohazard gear
  SALT No adverse events
Arm/Group | DL & Standard Clothing | DL & Biohazard Gear | Glidescope & Standard Clothing | Glidescope & Biohazard Gear | SALT & Standard Clothing | SALT and Biohazard Gear
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/37 | 0/37 | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/37 | 0/37 | 0/37 | 0/37

LIMITATIONS AND CAVEATS:
Limitations described in associated reference

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No